CLINICAL TRIAL: NCT06511362
Title: Comparative Effects of Perturbation and Functional Stabilization Training on Pain, Balance and Performance in Athletes With Patellofemoral Pain Syndrome
Brief Title: Comparative Effects of Perturbation and Functional Stabilization Training on Patellofemoral Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0478
Record Dates: First submitted 2024-06-11; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Anterior knee pain syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional stabilization training (Group 1)) (Experimental): The participants will perform Lateral bridge and ventral bridge(6 weeks protocol,5 sets 30 sec, 5 sec hold of each rep), Isometric hip abduction/lateral rotation in standing (first 2 weeks 2 sets 20 reps), Hip abduction/lateral rotation/extension in sidelying ( 6 week 2 sets 20 reps), Hip abduction/lateral rotation with slight knee and hip flexion in sidelying ( 6 week , 2 sets , 20 reps), Pelvic drop in standing ( 6 weeks , 3 sets 12 reps ) Hip lateral rotation in closed kinetic chain ( 6 weeks, 3 sets , 12 reps ) Single-leg deadlift (6-8 weeks , 3 sets , 12 reps) Single-leg squat ( last 2 weeks ,3 sets 12 reps) Prone knee flexion (6 weeks 2-3 sets , 12 reps) Seated knee extension (90°-45° of knee flexion)( 6 weeks ,2-3 sets 12 reps ) Single-leg standing on unstable platform ( 3 sets)
  Interventions: Procedure: Functional stabilization training
- Perturbation training(Group 2) (Experimental): Perform perturbation exercises that involve double leg foam balance activity (30-second hold), tilt board balance training (30-second hold), and roller board (30-second hold).
  Interventions: Procedure: perturbation exercises

INTERVENTIONS:
Procedure: Functional stabilization training — At the start of the study, a formal education session, lasting about 30 minutes will be given. whole treatment plan will be given for 8 weeks. Pre and post intervention measurements will be taken by using measuring tools.
  Arms: Functional stabilization training (Group 1))
Procedure: perturbation exercises — At the start of the study, a formal education session, lasting about 30 minutes will be given. whole treatment plan will be given for 8 weeks. Pre and post intervention measurements will be taken by using measuring tools.
  Arms: Perturbation training(Group 2)

SUMMARY:
The main objective of this study is to determine the comparative effects of perturbation and functional stabilization training on pain, balance, and performance in athletes with patellofemoral pain syndrome(PFPS). Patellofemoral pain syndrome is one of the well known causes of anterior knee joint pain. Proximal and distal joint muscle imbalances are the most predisposing factors in knee pain especially knee cap. Anterior knee pain Increase during flexion of the knee, i.e., jumping, running, squatting and descending stairs. PFPS have a crucial impact on balance and functional activities, particularly for young athletes under the age 40. Individuals with PFPS manifest abnormalities in the dynamic and kinematic balance of the lower extremity. Participants between the age of 18-30 with knee pain and have difficulty performing the activities. Perturbation training is the part of the neuromuscular training program include the balancing activities that test the balance during the rehabilitation program. Functional stabilization training is used to improve the muscle control and strength. This particular program focuses on improving balance and determining the effect of training on prformance and balance of athletes with PFPS.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome is one of the best-known causes of anterior knee joint pain. Proximal and distal joint muscle imbalances are the most prevalent factors in knee pain, especially in the knee cap. Patellofemoral pain syndrome is the most prevalent reason that brings young individuals to sports clinics. Possible mechanism that is used to explain the possibility of the occurrence of PFPS has been identified as joint pain, which in turn causes reflexive inhibition of VMO, Glut max, muscular weakness, reduces knee function, and causes discomfort and pain in the knee joint. Pain is aggravated with repetitive activities such as squatting, descending stairs, running and jumping. Individuals with PFPS may experience a loss of equilibrium and impaired function due to a lack of proprioception. Neuromuscular electrical stimulation, hip abductors and external rotator strengthening with proprioceptive training, and mayofascial release to the gluteal medius are some of the techniques that can be used for the management of PFPS. Athletic performance depends on the number of skills that require balance and muscular control. This particular study focuses on the comparative effects of functional stabilization and perturbation training.

A randomized clinical study will be conducted at pakistan sports board Board in Lahore on athletes with patellofemoral pain syndrome. The sample size of the study was calculated using G.Power. Non -Probability convenient sampling technique will be used for research. The sample size will be 34. The sample will be split into 2 groups. FSE along with traditional treatment, will be given to Group 1 and perturbation training will be given to Group 2. Tools that will be used to assess the baseline measures include (NPRS), horizontal and vertical jump tests, the lower extremity functional scale (LEFS), 40-yard splint tests, and the star excursion balance test before and after the intervention. The data will be analyzed using SPSS version 25. First, the Shapiro-Wilk test will be used to determine the normality of the data; the P-value will be greater than 0.05, and the data will be distributed normally. After assessing the normality of the data, it will be decided whether a parametric or non-parametric test will be used withn and between two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Anterior knee pain.
2. Age between 15 to 30.
3. Pain between 3 to 10 on NPRS.

Exclusion Criteria:

1. patellar fracture.
2. Intra-articular pathology( ligamental and meniscal injury of the knee).
3. Knee surgery
4. Fracture of hip, knee, shin bone and foot
5. Vestibular and visual disorders

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — female athlete between the age of 15-30, having with knee pain.
Enrollment: 26 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-25 (Estimated)

PRIMARY OUTCOMES:
A numerical pain rating scale | 10 months
  this numeric pain rating scale will use to assess the level of pain. This scale consist of values from 0 to 10. 0 represent to no pain where as 10 indicate to worst pain. Scale is subdivided into 3 level. Level 1 range from 0 to 3 interpret mild pain. Level 2 having range from 4 to 6 interpret individual has moderate pain and level 3 have value from 7 to 10 indicate the severe pain.
horizontal jump test (meters) | 10 months
  This test will be used to assess the performance of athletes. Participants must stand with their toes behind the zero-centimeter mark with the tape measure and jump as far as they can with two feet with swinging arms and bending knees. In this test, the participant must land a stick and measure the distance from the takeoff to the contact point after jumping. This scale is rated as excellent if a female athlete covers a distance >1.91 meters; 1.90-1.71 meters indicates above average; 1.70-1.60 meters indicates average; distances between 1.59 and 1.47 meters indicate below average; and distances covered by the athlete <1.47 meters represent poor distance or performance.
vertical jumps tests(cm) | 10 months
  Vertical jump test use to assess the performance of athlete(lower extremity strength). To perform this test athlete warm up for 10 minutes. Then, they perform this test by standing side onto the wall. Participants reach as high as possible with one hand mark as M1 after that they jump as high as possible, which mark as M2. Measure the distance between M1and M2. Distance measure in cm. The distance >60 cm consider as excellent, between 46-60 cm consider as above average, between 31-45 cm consider as average, 21-30 cm consider as below average and distance <20 cm consider as poor performance(strength)
40-yard sprint test (sec) | 10 months
  This test is used to assess speed, agility, and quickness. In this test, mark a 40-yard distance on the floor. Athletes run from the starting point to the finishing point. The time in seconds was measured by using a stopwatch to cover the 40-yard (36.6-meter) distance.
lower extremity functional scale | 10 months
  This test is used as a performance assessment tool. This test consists of 20 questions relating to the person's ability to perform tasks related to daily life. A scoring system is available to predict the functional level. 0-20 scores represent severe functional limitations. 21-40 scores indicate moderate functional limitation; 41-60 scores show mild functional limitation; and 61-80 scores show minimum and no functional limitation.
star excursion balance test(cm) | 10 months
  The star excursion balance test (SEBT) is described as a tool to assess the dynamic balance. Draw a star shape with tape on the floor, separated by a 45-degree angle. It involves reaching in multiple directions, mostly eight, while maintaining balance on one leg. Anterior, anteromedial, lateral, anterolateral, medial, posteromedial, posterior, and posteromedial are the eight directions. Relative distance percentage in each direction is measured by using the formula average distance in one direction/leg length*100. The average distance is measured by taking 3 readings of distance in each direction and dividing by 3.Reading must be done with both the right and left legs.

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, T-DPT, Principal Investigator — Riphah inernational university.
Locations (1):
- Pakistan sports board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available to other researcher